CLINICAL TRIAL: NCT02603445
Title: A Phase Ib Dose Escalation Study of BCL201 in Combination With Idelalisib in Patients With Follicular Lymphoma (FL) and Mantle Cell Lymphoma (MCL)
Brief Title: Study of Safety and Efficacy of BCL201 and Idelalisib in Patients With FL and MCL
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CBCL201X2102C
Record Dates: First submitted 2015-10-08; First posted 2015-11-11 (Estimated); Last update posted 2020-02-24 (Actual); Status verified 2020-02

CONDITIONS: Follicular Lymphoma, Mantle Cell Lymphoma
Keywords: BCL201; idelalisib; Follicular lymphoma; FL; mantle cell lymphoma; MCL
MeSH Terms: conditions — Lymphoma, Follicular; Lymphoma, Mantle-Cell | interventions — S55746; idelalisib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Follicular lymphoma (FL) (Experimental)
  Interventions: Drug: BCL201; Drug: Idelalisib
- Mantle cell lymphoma (MCL) (Experimental)
  Interventions: Drug: BCL201; Drug: Idelalisib

INTERVENTIONS:
Drug: BCL201
  Other Names: S55746
Drug: Idelalisib
  Other Names: Idela

SUMMARY:
This is a phase Ib multi-center, open-label study: escalation part followed by expansion part. The primary purpose of the Phase Ib CBCL201X2102C study is to characterize the safety and tolerability of BCL201 combined with idelalisib in patients with FL and MCL.

Approximately 65 patients are to be enrolled.

The primary endpoint for the Phase Ib is frequency, severity and seriousness of AEs, lab abnormalities and other safety parameters such as ECG changes. An adaptive Bayesian logistic regression model (BLRM) will guide the dose escalation to determine the MTD/RDE in phase Ib. In addition Bayesian regression models will be used to estimate the dose-exposure relationships for both BCL201 and idelalisib in order to guide the escalation steps. A Bayesian method for the expansion part will be used for the primary activity objective.

The study data will be analyzed and reported based on all patients' data of the escalation and expansion part.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed diagnosis of FL or MCL according to WHO 2008
* Relapsed or refractory with at least one (FL) or two (MCL), but not more than four, prior lines of antineoplastic regimens.
* Either FDG-avid on FDG-PET or measurable disease by CT on cross sectional imaging: > 1.5 cm for nodal lesion, > 1.0 cm for extra nodal lesion.
* Eastern Cooperative Oncology Group (ECOG) performance status of ≤ 2

Exclusion Criteria:

* For dose escalation part: Patients with MCL at high risk for tumor lysis syndrome
* Prior treatment with PI3Kδ or Bcl-2 inhibitors.
* Any other malignant disease
* History of serious allergic reactions including anaphylaxis and toxic epidermal necrolysis
* Inadequate organ function
* Concomitant treatment with:
* Strong CYP3A4/5 inducers or inhibitors
* Sensitive CYP3A4/5 substrates or CYP3A4/5 substrates with narrow therapeutic index (NTI)
* Sensitive CYP2D6 substrates or CYP2D6 substrates with NTI
* Selected dual substrates of CYP3A4/5 and CYP2C8
* Selected dual substrates of CYP3A4/5 and CYP2D6
* Selected dual substrates of OATP and CYP450
* Selected dual substrates of CYP3A4/5 and P-gp
* NTI P-gp substrates
* QT prolonging drugs with a known risk to induce TdP
* Proton pump inhibitors
* Treatment by warfarin or equivalent vitamin K antagonists.
* Other investigational therapies
* Herbal preparations/ medications
* Grapefruit, Seville oranges or products containing either juice

Other protocol-defined inclusion/exclusion may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2015-11-16 (Actual); Primary Completion 2018-07-10 (Actual); Study Completion 2018-07-10 (Actual)

PRIMARY OUTCOMES:
Number of participants with adverse events (AEs) | 24 months
  Characterized by Frequency, severity and seriousness of AEs, lab abnormalities and other safety parameters such as electrocardiogram (ECG) changes

SECONDARY OUTCOMES:
Incidence rate of dose limiting toxicities (DLTs) | 24 months
Exposure to BCL201 and idelalisib as measured by AUC0-24h at C1D15 | Cycle = 28 days
Plasma concentration of BCL201, idelalisib and GS-563117 (metabolite of idelalisib) | 24 Months
AUC pharmacokinetics (PK) parameter for BCL201, idelalisib and GS-563117 | 24 months
Objective Response Rate (ORR) | 24 months
Best Overall Response (BOR) | 24 months
Duration of Response (DOR) | 24 months
Complete Response (CR) | 24 months
Partial Response (PR) | 24 months
Stable disease (SD) | 24 months
Cmax pharmacokinetics (PK) parameter for BCL201, idelalisib and GS-563117 | 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (7):
- United States (2):
  - Novartis Investigative Site, New York, New York
  - Novartis Investigative Site, Houston, Texas
- Novartis Investigative Site, Salzburg, Austria
- France (2):
  - Novartis Investigative Site, Pierre-Bénite
  - Novartis Investigative Site, Toulouse
- Germany (2):
  - Novartis Investigative Site, Freiburg im Breisgau
  - Novartis Investigative Site, Mainz

IPD SHARING:
Plan to Share IPD: No